CLINICAL TRIAL: NCT02094105
Title: Effect of Endoscopic Screening on Esophageal Cancer Incidence and Mortality: 10-year Follow up of a Community-based, Controlled Study Among High Risk Population in China
Brief Title: Endoscopic Screening on Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Youlin Qiao, Professor and Director of Department of Cancer Epidemiology, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ESCC01
Record Dates: First submitted 2014-03-20; First posted 2014-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal cancer; screening; endoscopy; prevention
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- screening (Experimental): endoscopy examination with iodine staining
  Interventions: Procedure: Endoscopy examination with iodine staining
- control (No Intervention): 1/10 sampling questionnaire interview for control group.

INTERVENTIONS:
Procedure: Endoscopy examination with iodine staining — Endoscopy examination with Lugol's iodine staining and questionnaire once time and early treatment on precancerous lesions was undergone for the intervention group.
  Arms: screening

SUMMARY:
Importance: There are no global screening recommendations for esophageal squamous cell carcinoma (ESCC). Endoscopic screening has been investigated in high incidence areas of China since 1970's. But up until now there no apparent evidence that would lead to a reduction in disease morbidity and mortality.

Objective: To evaluate whether endoscopic screening and early intervention program could reduce the incidence or mortality of ESCC.

Design: Community-based, controlled cohort study among 45 386 residents, Endoscopy screening was completed from November 1999 to May of 2000. Subjects in intervention group were examined once during intervention period. The study follow-up concluded in December 2009.

Setting: High risk area of ESCC in China

Participants:Cluster sampling from communities with high rates of esophageal cancer. A set of villages with was selected as the study intervention community. Age 40 to 69 years residents were selected as an eligible population. Another set of villages was select as the control population. Buffer villages were set up between intervention and control group.

Intervention: Endoscopy with Lugol's iodine staining and early treatment on precancerous lesions was undergone for the intervention group.

Main Outcome(s) and Measure(s): Incidence and mortality ESCC

ELIGIBILITY:
Inclusion Criteria:

* local residents
* Men and women aged 40 to 69 years
* no contraindications for endoscopic examinations (e.g. history of reaction of iodine or lidocaine), and who were mentally and physically competent to provide written informed consent.
* informed consent

Exclusion Criteria:

* Not local residents
* age younger than 40 yrs and older than 69 yrs
* History of reaction of iodine or lidocaine
* contraindications for endoscopic examinations

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45386 (Actual)
Dates: Start 1999-11; Primary Completion 2009-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
incidence and mortality of ESCC | 10 years

SECONDARY OUTCOMES:
Cumulative incidence and mortality of total cancer, and gastric cardia cancer | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Youlin Qiao, PhD, Principal Investigator — Department of Cancer Epidemiology, Cancer Institute, Chinese Academy of Medical Sciences, & Peking Union Medical College
Locations (1):
- Cancer Institute/Hospital of Ci County, Handan, Hebei, China

REFERENCES:
- [Background] Drahos J, Wu M, Anderson WF, Trivers KF, King J, Rosenberg PS, Eheman C, Cook MB. Regional variations in esophageal cancer rates by census region in the United States, 1999-2008. PLoS One. 2013 Jul 4;8(7):e67913. doi: 10.1371/journal.pone.0067913. Print 2013. PMID 23861830
- [Background] Gonzalez L, Magno P, Ortiz AP, Ortiz-Ortiz K, Hess K, Nogueras-Gonzalez GM, Suarez E. Esophageal cancer incidence rates by histological type and overall: Puerto Rico versus the United States Surveillance, Epidemiology, and End Results population, 1992-2005. Cancer Epidemiol. 2013 Feb;37(1):5-10. doi: 10.1016/j.canep.2012.09.002. Epub 2012 Oct 11. PMID 23063415
- [Background] Cook MB, Chow WH, Devesa SS. Oesophageal cancer incidence in the United States by race, sex, and histologic type, 1977-2005. Br J Cancer. 2009 Sep 1;101(5):855-9. doi: 10.1038/sj.bjc.6605246. Epub 2009 Aug 11. PMID 19672254
- [Background] Cohen AM, Konigsberg IR. A clonal approach to the problem of neural crest determination. Dev Biol. 1975 Oct;46(2):262-80. doi: 10.1016/0012-1606(75)90104-9. No abstract available. PMID 1183721
- [Background] Wei WQ, Yang J, Zhang SW, Chen WQ, Qiao YL. [Analysis of the esophageal cancer mortality in 2004 - 2005 and its trends during last 30 years in China]. Zhonghua Yu Fang Yi Xue Za Zhi. 2010 May;44(5):398-402. Chinese. PMID 20654227
- [Background] Hiripi E, Jansen L, Gondos A, Emrich K, Holleczek B, Katalinic A, Luttmann S, Nennecke A, Brenner H; Gekid Cancer Survival Working Group. Survival of stomach and esophagus cancer patients in Germany in the early 21st century. Acta Oncol. 2012 Sep;51(7):906-14. doi: 10.3109/0284186X.2012.673732. Epub 2012 Apr 23. PMID 22524212